CLINICAL TRIAL: NCT00903578
Title: Impact of FGF-23 and Serum Phosphate on Allograft Function and Mortality in Kidney Allograft Recipients
Brief Title: Impact of Fibroblast Growth Factor 23 (FGF-23) and Serum Phosphate on Allograft Function and Mortality in Kidney Allograft Recipients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Sinee Disthabanchong, M.D, Ramathibodi Hospital, Mahidol University
Other Study IDs: KT-1
Record Dates: First submitted 2009-05-01; First posted 2009-05-18 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Kidney Transplantation
Keywords: FGF-23; vitamin D; phosphate; allograft dysfunction; mortality

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kidney transplant recipients

SUMMARY:
The present study will examine whether serum FGF-23 and serum phosphate at baseline of kidney transplant recipients can predict progression of allograft dysfunction at 3 years and all-cause mortality at 5 years.

ELIGIBILITY:
Inclusion Criteria:

* at least one year post-transplantation
* no more than 10% increase in serum creatinine for the past 3 months

Exclusion Criteria:

* refuse to participate in the study
* any acute illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-05; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Progression of allograft dysfunction and all-cause Mortality | 3 and 5 years

SECONDARY OUTCOMES:
Relationship of FGF-23 and 25-OH-D, 1-25-OH-D, PTH, calcium, phosphate, urine phosphate and eGFR | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sinee Disthabanchong, M.D., Principal Investigator — Ramathibodi Hospital, Mahidol University
Locations (1):
- Ramathibodi Hospital, Mahidol University, Phayathai, Bangkok, Thailand